CLINICAL TRIAL: NCT01577355
Title: Disposition of [14C]-LY2784544 Following Oral Administration in Healthy Male Subjects
Brief Title: A Study of LY2784544 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14484; I3X-MC-JHTD (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-04-11; First posted 2012-04-13 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-07

CONDITIONS: Healthy Male Volunteers
MeSH Terms: interventions — Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [C14]-LY2784544 (Experimental): Single 30 mg oral dose containing 100 micro curies of LY2784544
  Interventions: Radiation: Drug

INTERVENTIONS:
Radiation: Drug — Single 30 mg oral dose containing 100 micro curies of LY2784544

SUMMARY:
This is a single dose study of radiolabelled LY2784544 in healthy male subjects to study the absorption, distribution, metabolism and excretion of LY2784544. This study is for research purposes only and is not intended to treat any medical condition.

DETAILED DESCRIPTION:
This study is approximately 10 days long, (minimum 5 days, maximum 15 days) not including screening or follow up. Screening is required within 28 days prior to the first dose of study drug and follow up is required at least 7 days after discharge from the clinical research unit.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy males as determined by medical history and physical examination

  * Will either be sterile or, if sexually active, agree to use a reliable method of birth control from the day before dosing until 3 months after the end of the study
* Have a body mass index (BMI) of 19 to 29 kg/m^2, inclusive
* Have clinical laboratory test results within the normal reference range for the Clinical Research Unit (CRU) or results with acceptable deviations which are judged to be not clinically significant by the investigator
* Normal blood pressure (BP) and heart rate (sitting) as determined by the investigator
* Have venous access sufficient to allow for blood sampling as per the study requirements
* Are reliable and willing to make themselves available for the duration of the study and are willing to abide by the CRU policies and procedures and study restrictions
* Have given written informed consent approved by Lilly and the institutional review board (IRB) governing the CRU

Exclusion Criteria:

* Are currently enrolled in, have completed, or discontinued within the last 30 days from a clinical study involving an investigational product or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have known allergies to LY2784544 or related compounds
* Have previously completed or withdrawn from this study or any other study investigating LY2784544
* Have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Have a history or evidence of significant active neuropsychiatric disease and in particular evidence of significant medical or psychiatric illness within the past 12 months or have suicidal risk at the time of screening in the opinion of the investigator
* Have any other condition that in the opinion of the investigator would preclude participation in the study
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Show evidence of hepatitis C and/or positive hepatitis C antibody
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen
* Use of herbal preparations containing St. John's Wort, kava, garlic, ginger, gingko biloba, or guarana within 14 days prior to admission or at any time during the study
* Intent to use over-the-counter (OTC) medication or prescription medication within 7 days prior to dosing or at any time during the study
* Consumption of grapefruit or grapefruit-containing foods or grapefruit-containing juices, Seville oranges or Seville orange juices, and star fruit or star fruit juices within 7 days prior to dosing or at any time during the study
* Have an average weekly alcohol intake that exceeds 21 units per week or are unwilling to stop alcohol consumption for the duration of the study
* Have donated blood of more than 500 mL within the last month
* Have participated in a [14C]-study within the last 6 months prior to admission for this study. The total exposure from this study and the previous study must be within the Code of Federal Regulations (CFR) recommended levels considered safe (per 21 CFR 361.1), less than 5000 millirems (mrem)/year whole body annual exposure
* Exposure to significant radiation within 12 months prior to dose (for example, serial X-ray or computed tomography scans, barium meal, current employment in a job requiring radiation exposure monitoring)
* Are currently smokers or users of tobacco or nicotine-replacement products within the 6 months prior to study entry
* Baseline 12-lead electrocardiogram (ECG) with a corrected QT (Bazett's) interval of >450 msec and/or have an abnormality in the 12-lead ECG that, in the opinion of the investigator, increases the risks associated with participating in the study
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Have a history of congestive heart failure, unstable angina, myocardial infarction, or documented history of ventricular arrhythmia
* Gastrointestinal disorders causing clinically significant symptoms such as nausea, vomiting, and diarrhea, or malabsorption syndromes
* Evidence of active renal disease (e.g., diabetic renal disease, polycystic kidney disease) or creatinine clearance (CrCl) less than 70 mL/min
* Urinalysis with ≥1+ protein or ≥1+ blood (unless attributable to an acute condition that is resolved prior to dosing)
* Use of drugs with narrow therapeutic windows and that are also known substrates of Cytochrome P450 (CYP)1A2, CYP2B6, and CYP3A are specifically excluded
* Use of antacids and proton pump inhibitors
* Typically do not produce at least one bowel movement per day

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2012-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Urinary and fecal excretion of LY2784544 radioactivity over time expressed as a percentage of the total radioactive dose administered | Predose up to 14 days post dose

SECONDARY OUTCOMES:
Plasma pharmacokinetics of LY2784544 and radioactivity maximum observed concentration (Cmax) | Predose up to 14 days post dose
Plasma pharmacokinetics of LY27854544 and radioactivity time of maximum observed concentration (tmax) | Predose up to 14 days post dose
Plasma pharmacokinetics of LY2784544 and radioactivity area under the concentration-time curve from time zero to the last timepoint with a measurable concentration (AUC 0 to tlast) | Predose up to 14 days post dose
Relative abundance of LY2784544 and the metabolites of LY2784544 in urine and feces | Predose up to 14 days post dose
Relative abundance of LY2784544 and the metabolites of LY2784544 in plasma | Predose up to 14 days post dose
Plasma pharmacokinetics of LY2784544 and radioactivity half-life | Predose up to 14 days postdose

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madison, Wisconsin, United States